CLINICAL TRIAL: NCT01477567
Title: A Single Ascending Dose (SAD) Study of LY3009385 in Healthy Volunteers
Brief Title: A First-in-Human Study of LY3009385 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 14195; I5O-FW-GTCA (Other: Eli Lilly and Company)
Record Dates: First submitted 2011-11-18; First posted 2011-11-22 (Estimated); Results first posted 2014-10-06 (Estimated); Last update posted 2014-10-06 (Estimated); Status verified 2014-10

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (7):
- 0.3 mg LY3009385 (Experimental): LY3009385: 0.3 milligrams (mg), subcutaneous (SC) injection, single dose on Day 1
  Interventions: Drug: LY3009385
- 1 mg LY3009385 (Experimental): LY3009385: 1 milligrams (mg), subcutaneous (SC) injection, single dose on Day 1
  Interventions: Drug: LY3009385
- 3 mg LY3009385 (Experimental): LY3009385: 3 milligrams (mg), subcutaneous (SC) injection, single dose on Day 1
  Interventions: Drug: LY3009385
- 9 mg LY3009385 (Experimental): LY3009385: 9 milligrams (mg), subcutaneous (SC) injection, single dose on Day 1
  Interventions: Drug: LY3009385
- 22 mg LY3009385 (Experimental): LY3009385: 22 milligrams (mg), subcutaneous (SC) injection, single dose on Day 1
  Interventions: Drug: LY3009385
- 54 mg LY3009385 (Experimental): LY3009385: 54 milligrams (mg), subcutaneous (SC) injection, single dose on Day 1
  Interventions: Drug: LY3009385
- Placebo (Placebo Comparator): Placebo: saline, subcutaneous (SC) injection, single dose on Day 1
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LY3009385
  Arms: 0.3 mg LY3009385; 1 mg LY3009385; 22 mg LY3009385; 3 mg LY3009385; 54 mg LY3009385; 9 mg LY3009385
Drug: Placebo
  Arms: Placebo

SUMMARY:
The main purpose of this study is to determine the safety of LY3009385 in healthy participants. The study drug is given as a single dose, by injections under the skin. Side effects will be documented. This study is approximately 28 days not including screening. Screening is required within 28 days prior to the start of the study.

DETAILED DESCRIPTION:
This is a single ascending dose study that examines the safety and tolerability, pharmacokinetics (PK), and pharmacodynamic (PD) effects of single doses of LY3009385 administered subcutaneously to healthy participants. The planned dose levels are 0.3, 1, 3, 9, 27, and 54 milligrams (mg). Within each dose level, participants are randomized to receive either LY3009385 or Placebo.

Adjustments to the dose levels were permitted after review of emerging safety, PK, and glycemic data.

The actual LY3009385 dose levels tested during this study were 0.3, 1, 3, 9, 22, and 54 mg.

ELIGIBILITY:
Inclusion Criteria:

* Are a healthy male or a female who cannot become pregnant
* Have a body mass index (BMI) of 18.5 to 32.0 kilograms per meter squared (kg/m^2) at screening
* Have blood pressure, pulse rate, as well as blood and urine laboratory test results acceptable for the study
* Have veins suitable for easy blood collection
* Are reliable and willing to be available for the whole study and be willing to follow study procedures
* Have given consent to participate in this study

Exclusion Criteria:

* Are currently participating in or were in another new drug or device or in any medical research study in the last 30 days
* Currently have or used to have allergies or other health problems or laboratory test results that in the opinion of the doctor, could make it unsafe for the participant to participate, or interfere with understanding the results of this study
* Have received live vaccine(s) within 1 month of screening, or intend to during the study
* Have received treatment with biologic agents (such as monoclonal antibodies) within 3 months or 5 half-lives (whichever is longer) prior to dosing
* Have a weakened immune system
* Have previously completed or withdrawn from this study
* Have illnesses or conditions that may increase risk when taking the study medication or interfere with the interpretation of data in this study
* Have electrocardiogram (ECG) readings that are not suitable for the study
* Are using or intend to use over-the-counter medications or prescription medications within 7 and 14 days (respectively) from the start of the first study dosing until end of the study
* Have a history of drug or alcohol abuse
* Are infected with hepatitis B
* Are infected with human immunodeficiency virus (HIV)
* Have donated 450 milliliters (mL) or more of blood in the last 3 months or made any blood donation within the last month
* Have a regular alcohol intake greater than 21 units per week (males) and 14 units per week (females) or are unwilling to abstain from alcohol 24 hours before dosing until the completion of each inpatient study period
* Smoke more than 10 cigarettes per day or are unable or unwilling to refrain from smoking while at the clinic
* Are unwilling or unable to follow dietary requirements/restrictions for the study and only consume only the meals provided during inpatient stays at the clinical research unit
* Are deemed unsuitable to participate by the study doctor for any other reasons

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Singapore, Singapore

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 0.3 mg LY3009385 | 1 mg LY3009385 | 3 mg LY3009385 | 9 mg LY3009385 | 22 mg LY3009385 | 54 mg LY3009385 | Placebo
Started | 5 | 6 | 6 | 6 | 6 | 5 | 6
Received at Least 1 Dose of Study Drug | 5 | 6 | 6 | 6 | 6 | 5 | 6
Completed | 5 | 6 | 6 | 6 | 6 | 5 | 6
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.3 mg LY3009385 | 1 mg LY3009385 | 3 mg LY3009385 | 9 mg LY3009385 | 22 mg LY3009385 | 54 mg LY3009385 | Placebo | Total
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5 | 6 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.2 (13.5) | 36.7 (12.5) | 33.3 (14.0) | 31.7 (8.4) | 34.7 (10.4) | 34.6 (9.9) | 27.5 (4.3) | 33.8 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Male | 5 | 6 | 6 | 5 | 5 | 5 | 6 | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 5 | 6 | 6 | 6 | 6 | 5 | 6 | 40
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 5 | 6 | 6 | 6 | 6 | 5 | 6 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Singapore | 5 | 6 | 6 | 6 | 6 | 5 | 6 | 40
Fasting Blood Glucose [Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)] | 82.84 (4.99) | 92.40 (4.86) | 84.45 (10.60) | 96.02 (8.35) | 89.40 (6.29) | 92.46 (11.12) | 89.08 (5.17) | 89.62 (8.29)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With One or More Drug-related Adverse Events (AEs) or Any Serious AEs
Description: The number of participants with 1 or more AEs assessed as related to the study drug and is summarized cumulatively. In addition, the number of participants with 1 or more serious AEs is summarized cumulatively. A serious AE is defined as an event that results in death, initial or prolonged hospitalization, is life-threatening, leads to persistent or significant disability/incapacity, is associated with congenital anomaly/birth defect, or is considered significant by the investigator for any other reason. A summary of serious and other non-serious adverse events regardless of causality is located in the Reported Adverse Events module.
Time Frame: Baseline through Day 28
Population: All enrolled participants.
Measure: Number; unit: participants
Arm/Group | 0.3 mg LY3009385 | 1 mg LY3009385 | 3 mg LY3009385 | 9 mg LY3009385 | 22 mg LY3009385 | 54 mg LY3009385 | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5 | 6
participants
  Study Drug-Related AEs | 1 | 1 | 1 | 2 | 5 | 5 | 2
  Serious AEs | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Pharmacokinetics: Area Under the Concentration Curve (AUC) of LY3009385
Description: LY3009385 exposure in terms of AUC from time 0 extrapolated to infinity (AUC[0-inf]) is summarized.
Time Frame: Predose through Day 28
Population: Participants who received a dose of LY3009385 and had sufficient quantifiable plasma LY3009385 concentrations in the terminal phase.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms times hours per milliliter
Arm/Group | 0.3 mg LY3009385 | 1 mg LY3009385 | 3 mg LY3009385 | 9 mg LY3009385 | 22 mg LY3009385 | 54 mg LY3009385
Number analyzed (Participants) | 3 | 6 | 6 | 6 | 6 | 4
micrograms times hours per milliliter | 4.81 (76) | 9.49 (213) | 53.1 (54) | 214 (42) | 757 (59) | 1670 (27)

3. Secondary Outcome: Pharmacokinetics: Maximum Concentration (Cmax)
Description: The maximum observed plasma concentration (Cmax) of LY3009385 is summarized.
Time Frame: Predose through Day 28
Population: Participants who received a dose of LY3009385 and had evaluable LY3009385 concentration data.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter
Arm/Group | 0.3 mg LY3009385 | 1 mg LY3009385 | 3 mg LY3009385 | 9 mg LY3009385 | 22 mg LY3009385 | 54 mg LY3009385
Number analyzed (Participants) | 4 | 6 | 6 | 6 | 6 | 5
nanograms per milliliter | 14.1 (41) | 51.9 (118) | 180 (46) | 847 (36) | 2030 (14) | 4810 (19)

4. Secondary Outcome: Change in Level of Blood Glucose Before and After a Standard Meal
Description: The effect of LY3009385 on postprandial blood glucose was evaluated. Change from baseline area under the glucose concentration-time curve from time 0 to 6 hours after participants started eating a standardized breakfast (mixed-meal tolerance test) was calculated and summarized by treatment arm.
Time Frame: Baseline, Day 5, and Day 14
Population: Participants who received a dose of LY3009385 or Placebo and had evaluable blood glucose concentration data.
Measure: Mean (Standard Deviation); unit: milligrams times hours per deciliter
Arm/Group | 0.3 mg LY3009385 | 1 mg LY3009385 | 3 mg LY3009385 | 9 mg LY3009385 | 22 mg LY3009385 | 54 mg LY3009385 | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5 | 6
milligrams times hours per deciliter
  Day 5 (n= 5, 6, 6, 6, 6, 5, 6) | 76.54 (56.51) | -45.35 (18.27) | -8.44 (45.83) | -14.50 (36.92) | -31.33 (38.43) | -108.93 (25.67) | 4.73 (30.43)
  Day 14 (n= 0, 0, 6, 6, 6, 5, 4) | NA (NA) — The effect of LY3009385 on postprandial glucose concentrations was not evaluated on Day 14 for this treatment arm. | NA (NA) — The effect of LY3009385 on postprandial glucose concentrations was not evaluated on Day 14 for this treatment arm. | 42.30 (33.69) | -60.57 (52.29) | 5.16 (38.48) | -129.75 (27.55) | -3.54 (54.72)

5. Secondary Outcome: Change in Level of C-peptide Before and After a Standard Meal
Description: The effect of LY3009385 on postprandial c-peptide was assessed. Change from baseline area under the c-peptide concentration-time curve from time 0 to 4 hours after participants started eating a standardized breakfast (mixed-meal tolerance test) was calculated and summarized by treatment arm.
Time Frame: Baseline, Day 5, and Day 14
Population: Participants who received a dose of LY3009385 or Placebo and had evaluable c-peptide concentration data.
Measure: Mean (Standard Deviation); unit: picomoles times hours per liter
Arm/Group | 0.3 mg LY3009385 | 1 mg LY3009385 | 3 mg LY3009385 | 9 mg LY3009385 | 22 mg LY3009385 | 54 mg LY3009385 | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5 | 6
picomoles times hours per liter
  Day 5 (n= 5, 6, 6, 6, 6, 5, 6) | 932.50 (2402.47) | 2235.08 (1204.19) | 982.50 (1104.62) | 1510.58 (1289.05) | 640.25 (1572.44) | -116.50 (1414.08) | 866.50 (1954.39)
  Day 14 (n= 0, 0, 6, 6, 6, 5, 4) | NA (NA) — The effect of LY3009385 on postprandial c-peptide levels was not evaluated on Day 14 for this treatment arm. | NA (NA) — The effect of LY3009385 on postprandial c-peptide levels was not evaluated on Day 14 for this treatment arm. | -363.92 (1174.13) | 1324.75 (2627.97) | 511.67 (786.06) | 955.40 (1463.97) | -959.13 (2164.81)

6. Secondary Outcome: Change in Level of Glucagon Before and After a Standard Meal
Description: The effect of LY3009385 on postprandial glucagon levels was assessed. Change from baseline glucagon concentrations 2 hours after participants started eating a standardized breakfast (mixed-meal tolerance test) were calculated and summarized by treatment arm.
Time Frame: Baseline, Day 14
Population: Participants who received a dose of LY3009385 or Placebo and have evaluable glucagon concentration data. The effect of LY3009385 on postprandial glucagon concentrations was not evaluated on Day 14 for the 0.3 and 1 mg treatment arms.
Measure: Mean (Standard Deviation); unit: picomoles per liter
Arm/Group | 3 mg LY3009385 | 9 mg LY3009385 | 22 mg LY3009385 | 54 mg LY3009385 | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 5 | 4
picomoles per liter | 0.93 (2.66) | -1.05 (2.59) | 0.68 (2.46) | 0.68 (2.52) | 0.48 (6.15)

7. Secondary Outcome: Number of Participants Forming Antibody to LY3009385
Description: The number of participants with postbaseline detection of LY3009385treatment-emergent (TE) antidrug antibodies (ADA), defined as a 4-fold increase in the ADA titer from baseline.
Time Frame: Baseline through Day 28
Population: Participants who received a dose of LY3009385 or Placebo.
Measure: Number; unit: participants
Arm/Group | 0.3 mg LY3009385 | 1 mg LY3009385 | 3 mg LY3009385 | 9 mg LY3009385 | 22 mg LY3009385 | 54 mg LY3009385 | Placebo
Number analyzed (Participants) | 5 | 6 | 6 | 6 | 6 | 5 | 6
participants | 1 | 2 | 2 | 2 | 2 | 0 | 0

ADVERSE EVENTS:
Groups:
- 1 mg LY3009385: LY3009385: 1 milligram (mg), subcutaneous (SC) injection, single dose on Day 1
Arm/Group | 0.3 mg LY3009385 | 1 mg LY3009385 | 3 mg LY3009385 | 9 mg LY3009385 | 22 mg LY3009385 | 54 mg LY3009385 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6 | 0/6 | 0/6 | 0/6 | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 5/5 | 6/6 | 6/6 | 5/6 | 6/6 | 5/5 | 5/6
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.3 mg LY3009385 (N=5) | 1 mg LY3009385 (N=6) | 3 mg LY3009385 (N=6) | 9 mg LY3009385 (N=6) | 22 mg LY3009385 (N=6) | 54 mg LY3009385 (N=5) | Placebo (N=6)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (5) | 0 (0)
Toothache (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 0 (0)
Application site erythema (General disorders) | 0 (0) | 4 (5) | 1 (1) | 2 (3) | 1 (2) | 2 (2) | 2 (2)
Application site pruritus (General disorders) | 0 (0) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 1 (1)
Application site rash (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Catheter site erythema (General disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 2 (3)
Catheter site haematoma (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Catheter site pain (General disorders) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hunger (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injection site haematoma (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vessel puncture site haematoma (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vessel puncture site thrombosis (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Procedural site reaction (Injury, poisoning and procedural complications) | 5 (10) | 2 (3) | 1 (1) | 3 (3) | 1 (3) | 1 (1) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 4 (5) | 1 (1)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 3 (3) | 5 (14) | 1 (1)
Increased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes